CLINICAL TRIAL: NCT01280045
Title: Influence of the Aromatase Inhibitor Anastrozole and GnRH Analog Goserelin Acetate as Preoperative Treatment of Vaginal Surgical Treatment of Uterine Leiomyoma: Analysis of Intra and Immediate/Late Postoperative Patterns
Brief Title: Influence of Aromatase Inhibitors and GnRH Analogs to Treat Uterine Leiomyoma by Vaginal Hysterectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No grant was received then we stopped the recruitment
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, LUIZ GUSTAVO OLIVEIRA BRITO, Assistant Physician, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMRPUSP-UROGIN-001
Record Dates: First submitted 2011-01-10; First posted 2011-01-20 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: UTERINE LEIOMYOMA
MeSH Terms: conditions — Myofibroma | interventions — Hysterectomy, Vaginal

STUDY DESIGN:
Intervention Model Description: We woudl be comparing aromatase inhibitors versus GnRH analogs
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AROMATASE INHIBITOR (Experimental): this would be compared before and after VAGINAL HYSTERECTOMY
  Interventions: Procedure: VAGINAL HYSTERECTOMY
- GNRH ANALOG (Active Comparator): this would be compared before and after VAGINAL HYSTERECTOMY
  Interventions: Procedure: VAGINAL HYSTERECTOMY

INTERVENTIONS:
Procedure: VAGINAL HYSTERECTOMY — GOSERELINE ACETATE 10.8 MG FOR THREE MONTHS; ANASTROZOL ACETATE FOR THREE MONTHS
  Other Names: None declared

SUMMARY:
The investigators aimed to assess if use of aromatase inhibitors could decrease volume of uterine leiomyoma and cause same percentage of adverse effects during its use compared to GnRH analogs.

DETAILED DESCRIPTION:
Uterine leiomyoma is the most prevalent benign gynecologic tumor in women. Standard treatment is surgical (hysterectomy or myomectomy), and depends of many variables. If these tumors are large, preoperative assessment with clinical treatment may be useful in order to decrease its volume, improve hematologic patterns and modify surgical approach (vaginal or abdominal). It is well know that GnRH analogs can cause these goals; however, aromatase inhibitors are new promising drugs which are being used for reducing uterine leiomyoma's volume and few observational studies have shown this fact. The investigators are aiming to compare both treatments in a randomized controlled trial and see if it both treatments are similar or not in decreasing uterine leiomyoma's volume, influencing operative time, blood loss during surgery.

ELIGIBILITY:
Inclusion Criteria:

* WOMEN OVER 40 YEARS, UTERINE VOLUME HIGHER THAN 300 ML, MINIMAL ANATOMIC CONDITIONS FOR VAGINAL SURGERY

Exclusion Criteria:

* ACTIVE GYNECOLOGIC MALIGNANCY

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Operative Time | Intra-operative
  Intra-operative time

SECONDARY OUTCOMES:
Uterine Leiomyoma Volume | 3 Months After Treatment, During Surgery
  Volume measured by ultrasound

REFERENCES:
- [Result] Parsanezhad ME, Azmoon M, Alborzi S, Rajaeefard A, Zarei A, Kazerooni T, Frank V, Schmidt EH. A randomized, controlled clinical trial comparing the effects of aromatase inhibitor (letrozole) and gonadotropin-releasing hormone agonist (triptorelin) on uterine leiomyoma volume and hormonal status. Fertil Steril. 2010 Jan;93(1):192-8. doi: 10.1016/j.fertnstert.2008.09.064. Epub 2009 Jan 9. PMID 19135657